CLINICAL TRIAL: NCT01456312
Title: A Multi Center, Phase IIIb Study to Evaluate the Efficacy of Response Guided Therapy Using Quantitative HBsAg Measurement in Patient With HBeAg Positive Chronic Hepatitis B:
Brief Title: HBsAg Related Response Guided Therapy
Acronym: S-RGT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Kwan Sik Lee, professor, Gangnam Severance Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25588
Record Dates: First submitted 2011-10-15; First posted 2011-10-20 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Hepatitis B, Chronic
Keywords: Peginterferon alfa 2a; Entecavir; Response Guided Therapy; Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- HBsAg quantification>20,000 IU/ml (Sham Comparator): stop peginterferon alfa 2a if patients reach HBsAg quantification>20,000 Iu/ml at 12w
  Interventions: Drug: Peginterferon alfa-2a
- HBsAg<=1500IU/ml (Sham Comparator): extend peginterferon alfa 2a until 48weeks
  Interventions: Drug: Peginterferon alfa-2a
- HBsAg >1500 <=20,000 IU/ML (Sham Comparator): add Entecavir for 12w with peginterferon alfa 2a then, extend peginterferon alfa 2a until 48w
  Interventions: Drug: Peginterferon alfa-2a; Drug: Entecavir

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Duration and combination
  Other Names: Pegasys
Drug: Entecavir — combination
  Other Names: Baraclude Tab
  Arms: HBsAg >1500 <=20,000 IU/ML

SUMMARY:
Primary objective: Compare Pegasys RGT overall response rate (i.e., HBeAg seroconversion rate) with Pegasys mono historical response rate at week 72 (48 week treatment with 24 week follow up)

Secondary objective :

* The changes of HBsAg titer

  * The rate of combined HBeAg seroconversion and HBV DNA < 300 copies/mL

    * The rate of serum HBV DNA < 300 copies/mL ⅳ. The rate of ALT normalization

      * The rate of HBsAg loss ⅵ. The rate of serum HBV DNA < 10,000 copies/mL

DETAILED DESCRIPTION:
After 12w treatment of Pegasys, depends on results of quantitative HBsAg test, Patients will be allocated to one of three groups.

* HBsAg >20,000 : study termination
* Group A :1,500<HBsAg≤ 20,000
* Group B : .HBsAg ≤ 1500 At week 48, according to HbeAg seroconversion, patients will be allocated to one of two sub-groups(A-1, A-2, B-1, B-2) Patients are seen for evaluation at treatment weeks 4,8,12,24,36,48. Post-treatment assessments will be performed at 4,12 and 24 week during off-treatment phase for the assessment of the primary and main secondary endpoints of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Positive HBsAg for more than 6 months, positive HBeAg, detectable HBV DNA(patients must have > 100,000 copies/ml as measured by PCR) and anti-HBs negative
3. Elevated serum ALT > 2ULN but ≤ 10 × ULN as determined by two abnormal values taken ≥ 14 days apart during the six months before the first dose of study drug with at least one of the determinations obtained ≤ 35 days prior to the first dose.

Exclusion Criteria:

1. Patients must not have received antiviral therapy for their chronic hepatitis B. Patients who are expected to need systemic antiviral therapy other than that provided by the study at any time during their participation in the study are also excluded. Exception: patients who have had less than 6 months treatment of NA(Nucleos(t)ide analog) and more than 1 year wash-out period for systemic antiviral therapy and negative results in the NA resistance test at baseline are not excluded.
2. Positive test at screening for HAV IgM Ab, HCV-RNA or HCV Ab, HDV Ab or HIV Ab.
3. Diagnosed hepatic cellular carcinoma
4. Any evidence of decompensated liver disease (Childs B-C)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-02 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
HBeAg seroconversion | 24 weeks post treatment follow up

SECONDARY OUTCOMES:
The changes of HBsAg titer | baseline and 24weeks post treatment follow up

CONTACTS AND LOCATIONS:
Overall Officials: Kwansik Lee, professor, Study Chair — Gangnam Severance Hospital
Locations (1):
- Shinchon Severance Hospital, Seoul, Seoul, South Korea